CLINICAL TRIAL: NCT03994315
Title: Exclusively Formula-Fed Infants Effectively Colonizing With B. Infantis EVC001 From Lacto-N-Tetraose Supplementation
Brief Title: The EFFECT Study: Probiotic and HMO Supplementation in Infants
Acronym: EFFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evolve BioSystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EV-8901
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Infant Gut Microbiome
MeSH Terms: interventions — lacto-N-neotetraose

STUDY DESIGN:
Intervention Model Description: This study is a single-center, prospective, randomized, open-label study of an infant probiotic (B. infantis EVC001) and a prebiotic supplement (LNT) in exclusively formula-fed infants. Nine subjects will be randomized (1:1:1) using sealed envelopes into three treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- B. infantis EVC001 + LNT (3 g/L then 8 g/L) (Experimental): Infants will receive a once-daily oral feeding of B. infantis EVC001 (8.0 x 10^9 CFU) mixed with infant formula for 28 consecutive days. Group 1 [B. infantis + LNT (3 g/L then 8 g/L)] will also receive two dose-escalated concentrations of the prebiotic supplement (LNT) mixed with their infant formula for every formula preparation during the 28-day supplementation period. They will receive a concentration of 3 g/L for 2 weeks followed by 8 g/L for the next 2 weeks, without a washout period in between.
  Interventions: Other: B. infantis EVC001; Other: Lacto-N-tetraose (LNT)
- B. infantis EVC001 + LNT (6 g/L then 12 g/L) (Experimental): Infants will receive a once-daily oral feeding of B. infantis EVC001 (8.0 x 10^9 CFU) mixed with infant formula for 28 consecutive days. Group 2 [B. infantis + LNT (6 g/L then 12 g/L)] will also receive two dose-escalated concentrations of the prebiotic supplement (LNT) mixed with their infant formula for every formula preparation during the 28-day supplementation period. They will receive a concentration of 6 g/L for 2 weeks followed by 12 g/L for the next 2 weeks, without a washout period in between.
  Interventions: Other: B. infantis EVC001; Other: Lacto-N-tetraose (LNT)
- B. infantis EVC001 alone (Active Comparator): Infants will receive a once-daily oral feeding of B. infantis EVC001 (8.0 x 10^9 CFU) mixed with infant formula for 28 consecutive days.
  Interventions: Other: B. infantis EVC001

INTERVENTIONS:
Other: B. infantis EVC001 — Bifidobacterium longum subspecies infantis strain EVC001, designated a "Foods for Special Dietary Use" (FSDU)
  Other Names: Evivo
Other: Lacto-N-tetraose (LNT) — LNT is a human milk oligosaccharide (HMO) found in human breast milk and is a selective prebiotic for B. infantis.
  Arms: B. infantis EVC001 + LNT (3 g/L then 8 g/L); B. infantis EVC001 + LNT (6 g/L then 12 g/L)

SUMMARY:
Lacto-N-tetraose (LNT) is a human milk oligosaccharide (HMO) present in human colostrum and milk. HMOs are largely undigestable and have no direct nutritive benefit to the infant, but act as a prebiotic substrate for beneficial bacteria (bifidobacteria, in particular) in the infant gut. Exclusively formula-fed infants lack HMOs in their diet in the absence of naturally occurring HMOs from breast milk. The proposed clinical study will evaluate the ability of a prebiotic supplement (LNT) to initiate intestinal colonization of a probiotic strain (B. infantis EVC001) in exclusively formula-fed infants. B. infantis EVC001 has been shown to be well-tolerated and safely consumed in breastfed infants. This study also aims to evaluate the safety and tolerability of LNT in different doses when consumed daily with B. infantis EVC001.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized, open-label study of an infant probiotic (B. infantis EVC001) and a prebiotic supplement (LNT) in exclusively formula-fed infants. Nine subjects will be enrolled into three treatment arms:

* Group 1: 8 x 10^9 CFU B. infantis + LNT (3 g/L then 8 g/L)
* Group 2: 8 x 10^9 CFU B. infantis + LNT (6 g/L then 12 g/L)
* Group 3: 8 x 10^9 CFU B. infantis alone Study staff will be unblinded to the treatment assignments. Infants in all groups will receive a once-daily oral feeding of B. infantis EVC001 (8.0 x 10^9 CFU) mixed with infant formula for 28 consecutive days. Two of the treatment groups (Group 1 & Group 2) will also receive two dose-escalated concentrations of the prebiotic supplement (LNT) mixed with their daily infant formula: Group 1 will receive a concentration of 3 g/L for 2 weeks followed by 8 g/L for the next 2 weeks. Group 2 will receive a concentration of 6 g/L for 2 weeks followed by 12 g/L for the next 2 weeks. Infants consuming the LNT will cross over to the higher dose without a washout period in between. All infants will be evaluated for an additional 2 weeks after cessation of the supplement(s). The total duration of the study will be approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Infant is between 0 and 60 days of life at the time of enrollment
2. Infant is exclusively formula-fed with caregiver intent to continue exclusive formula feeding for the duration of the study (at least 7 weeks)
3. Infant is consuming cow's milk-based formula without probiotics
4. Term infant, born >37 weeks gestation
5. Infant is healthy and without medical complications
6. Infant's caregivers are willing to refrain from feeding their infant breast milk, solid foods, and non-study probiotics prior to study completion

Exclusion Criteria:

1. Infant was born with medical complications such as respiratory distress syndrome or birth defects
2. Infant has any gastrointestinal tract abnormalities
3. Infant has been diagnosed with failure to thrive
4. Infant has taken oral or IV antibiotics or antifungals within 4 weeks of enrollment or during the Lead-in Period
5. Infant is consuming partially hydrolyzed or extensively hydrolyzed infant formula because of gastrointestinal disturbance or gassiness/fussiness
6. Infant has consumed any breast milk within 7 days of enrollment or during the Lead-in Period
7. Infant has consumed any probiotics containing B. infantis since birth
8. Infant has consumed any Bifidobacterium-containing probiotics within 2 weeks of enrollment or during the Lead-in Period
9. Infant's caregivers plan to feed them any breast milk, solid foods, or non-study probiotics at any time throughout the duration of the study
10. Infant was born in a multiple birth
11. Infant lives in more than one location
12. Any infant who the investigator feels is not an appropriate study participant

Max Age: 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
B. infantis levels in infant stool | Baseline, Days 1-35, Day 40
  To evaluate the ability of different doses of a prebiotic supplement (LNT) to initiate intestinal colonization of a probiotic strain (B. infantis EVC001) in exclusively formula-fed infants. DNA will be extracted from stool swab samples and will be used for quantitative PCR to determine levels of B. infantis.

SECONDARY OUTCOMES:
Total infant gut microbiome modulation | Baseline, Days 5, 12, 19, 26, 40
  To evaluate the total gut microbiome modulation from supplementation of B. infantis with and without a prebiotic supplement (LNT) in exclusively formula-fed infants. DNA and RNA will be extracted from stool swab samples and will be used for next generation sequencing to determine relative abundance of the most abundant bacterial taxa.
Frequency of adverse events | During supplementation (Day 1 to Day 28) and Post-supplementation (Day 29 to Day 42)
  Frequency of treatment emergent adverse events (TEAEs), serious TEAEs and TEAEs causing premature discontinuation will be provided by treatment group.
Frequency of gastrointestinal symptoms warranting a doctor's visit | During supplementation (Day 1 to Day 28) and Post-supplementation (Day 29 to Day 42)
  Frequency of gastrointestinal symptoms warranting a doctor's visit will be provided by treatment group.
Frequency of adverse events resulting in withholding or discontinuing the study products | During supplementation (Day 1 to Day 28)
  Frequency of adverse events resulting in withholding or discontinuing the study products will be provided by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Rimon Youssef, MD, Principal Investigator — Coastal Pediatric Research
Locations (1):
- Coastal Pediatric Research, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No